CLINICAL TRIAL: NCT03501030
Title: Activity Restriction for Women With Arrested Preterm Labor: a Randomized Controlled Trial
Brief Title: Activity Restriction for Women With Arrested Preterm Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 29/18
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Single center, parallel group non-blinded, prospective, interventional non-pharmacologic, no profit, randomized and controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity restriction (Experimental): Women in the intervention group will be recommended activity restriction. Activity restriction is defined as the following forms of activity restriction: pelvic rest and prohibition of sexual activity, reduction of work and/or non work activity. Bed rest will not recommended.
  Interventions: Behavioral: Activity restriction
- No activity restriction (No Intervention): Women in the control group will not receive any reccomandation regarding activity restriction. Bed rest and abstain from sexual intercourse will also not recommended.

INTERVENTIONS:
Behavioral: Activity restriction — Women in the intervention group will be recommended activity restriction. Activity restriction is defined as the following forms of activity restriction: pelvic rest and prohibition of sexual activity, reduction of work and/or non work activity. Bed rest will not recommended.
  Arms: Activity restriction

SUMMARY:
to test the hypothesis that activity restriction in women with singleton gestations and with arrested PTL would reduce the rate of PTB.

DETAILED DESCRIPTION:
Preterm birth (PTB) is a major cause of perinatal morbidity and mortality. Worldwide, about 15 million babies are born too soon every year, causing 1.1 million deaths, as well as short- and long-term disability in countless survivors.

Preterm labor (PTL) is the final pathway for about 50% of all PTB. Tocolytic agents are drugs that can slow or stop labor contractions in the attempt to delay births preceded by PTL. Primary tocolysis is defined as tocolysis given on initial presentation of women with PTL. In most of these women, PTL stops, but as their risk of PTB remains high, some have advocated use of maintenance tocolysis, i.e. tocolysis after arrested PTL. So far, no maintenance tocolytic agent has been shown to be beneficial in preventing PTB.

Some authors have also advocated the use of activity restriction in women with arrested PTL to reduce the risk of PTB. Activity restriction is defined as the following forms of activity restriction: pelvic rest and prohibition of sexual activity, reduction of work and/or non work activity. So far, the benefit of activity restriction in women with arrested PTL is still subject of debate and no Randomized Controlled Trial (RCT) has been undertaken.

Thus, the aim of this trial is to test the hypothesis that activity restriction in women with singleton gestations and with arrested PTL would reduce the rate of PTB.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestations;
* arrested PTL;
* TVU CL < 25 mm;
* 18 years to 50 years.

Exclusion Criteria:

* multiple gestations;
* symptoms of PTL (not arrested PTL);
* TVU CL ≥ 25mm;
* premature rupture of amnion and chorion membranes (PROM) at the time of randomization;
* cerclage in situ at the time of randomization;
* pessary in situ at the time of randomization;
* vaginal bleeding at the time of randomization;
* women who are unconscious, severly ill, mentally handicapped;
* women under the age of 18 years or over the age of 50 years.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only pregnant women (limit to Female)
Enrollment: 120 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Preterm birth | 37 weeks of gestation
  Preterm delivery at less than 37 weeks of gestation

SECONDARY OUTCOMES:
Mean gestational age at delivery in weeks | At the time of delivery
  Mean gestational age at delivery in weeks
Mean latency | from randomization to delivery
  from randomization to delivery
admission to nicu | at the time of delivery until 28 days of life
  number of babies admitted to neonatal intensive care unit
neonatal death | at the time of delivery until 28 days of life
  death of a live-born baby
a composite of adverse perinatal outcome | at the time of delivery until 28 days of life
  defined as at least one of the following:
  * necrotizing enterocolitis (NEC);
  * intraventricular hemorrhage (IVH) grade 3 or higher;
  * respiratory distress syndrome (RDS);
  * bronchopulmonry dysplasia (BPD);
  * retinopathy of prematurity (ROP) requiring therapy;
  * blood-culture proven sepsis;
  * admission to neonatal intensive care unit (NICU);
  * neonatal death;
chorioamnionitis | at the time of delivery
  diagnosis of choriamnionitis at histological examination of the placenta.

CONTACTS AND LOCATIONS:
Locations (1):
- Giuseppe De Placido, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saccone G, Della Corte L, Cuomo L, Reppuccia S, Murolo C, Napoli FD, Locci M, Bifulco G. Activity restriction for women with arrested preterm labor: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Aug;5(8):100954. doi: 10.1016/j.ajogmf.2023.100954. Epub 2023 Apr 18. PMID 37080296